CLINICAL TRIAL: NCT02402127
Title: Evaluation of the Lubricity of Daily Disposable Silicone Hydrogel Contact Lenses After Wear
Brief Title: Lubricity Post-Wear - Competitive Lenses Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CLT567-P001
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Results first posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-07

CONDITIONS: Refractive Error
Keywords: Contact lenses; Lubricity
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- TruEye, MyDay, clariti 1day (Other): Narafilcon A contact lenses in Period 1, followed by stenfilcon A contact lenses in Period 2 and somofilcon A contact lenses in Period 3. Each product worn bilaterally (in both eyes) for 1 day (16 hours).
  Interventions: Device: Narafilcon A contact lenses; Device: Stenfilcon A contact lenses; Device: Somofilcon A contact lenses
- TruEye, clariti 1day, MyDay (Other): Narafilcon A contact lenses in Period 1, followed by somofilcon A contact lenses in Period 2 and stenfilcon A contact lenses in Period 3. Each product worn bilaterally for 1 day (16 hours).
  Interventions: Device: Narafilcon A contact lenses; Device: Stenfilcon A contact lenses; Device: Somofilcon A contact lenses
- MyDay, TruEye, clariti 1day (Other): Stenfilcon A contact lenses in Period 1, followed by narafilcon A contact lenses in Period 2 and somofilcon A contact lenses in Period 3. Each product worn bilaterally for 1 day (16 hours).
  Interventions: Device: Narafilcon A contact lenses; Device: Stenfilcon A contact lenses; Device: Somofilcon A contact lenses
- MyDay, clariti 1day, TruEye (Other): Stenfilcon A contact lenses in Period 1, followed by somofilcon A contact lenses in Period 2 and narafilcon A contact lenses in Period 3. Each product worn bilaterally for 1 day (16 hours).
  Interventions: Device: Narafilcon A contact lenses; Device: Stenfilcon A contact lenses; Device: Somofilcon A contact lenses
- Clariti 1day, TruEye, MyDay (Other): Somofilcon A contact lenses in Period 1, followed by narafilcon A contact lenses in Period 2 and stenfilcon A contact lenses in Period 3. Each product worn bilaterally for 1 day (16 hours).
  Interventions: Device: Narafilcon A contact lenses; Device: Stenfilcon A contact lenses; Device: Somofilcon A contact lenses
- Clariti 1day, MyDay, TruEye (Other): Somofilcon A contact lenses in Period 1, followed by stenfilcon A contact lenses in Period 2 and narafilcon A contact lenses in Period 3. Each product worn bilaterally for 1 day (16 hours).
  Interventions: Device: Narafilcon A contact lenses; Device: Stenfilcon A contact lenses; Device: Somofilcon A contact lenses

INTERVENTIONS:
Device: Narafilcon A contact lenses — Silicone hydrogel contact lenses for daily disposable wear
  Other Names: 1-DAY ACUVUE® TruEye® (TruEye)
Device: Stenfilcon A contact lenses — Silicone hydrogel contact lenses for daily disposable wear
  Other Names: MyDay™
Device: Somofilcon A contact lenses — Silicone hydrogel contact lenses for daily disposable wear
  Other Names: clariti® 1day

SUMMARY:
The purpose of this study is to measure the coefficient of friction of three silicone hydrogel, daily disposable contact lenses after 16 hours of wear.

DETAILED DESCRIPTION:
In this 3-treatment, 3-period, 6-sequence crossover study, each participant will wear all 3 products in randomized order, 1 product at a time, with a washout period of up to 7 days between treatment periods. Lenses will be collected for ex-vivo lubricity analysis. The ex-vivo lubricity analysis will be conducted under a separate non-clinical protocol.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form.
* Soft contact lens wearer (both eyes).
* Willing to wear study lenses at least 16 waking hours and attend all study visits.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear.
* Use of systemic or ocular medications for which contact lens wear could be contraindicated.
* Use of artificial tears and rewetting drops during the study.
* Monocular (only 1 eye with functional vision) or fit with only 1 lens.
* History of herpetic keratitis, ocular surgery, or irregular cornea.
* Pregnant.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Vision Care, Global Medical Affairs, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three investigational centers located in the United States.
Pre-assignment Details: All enrolled participants (24)
Groups:
- TruEye, MyDay, Clariti 1day: Narafilcon A contact lenses in Period 1, followed by stenfilcon A contact lenses in Period 2 and somofilcon A contact lenses in Period 3
- TruEye, Clariti 1day, MyDay: Narafilcon A contact lenses in Period 1, followed by somofilcon A contact lenses in Period 2 and stenfilcon A contact lenses in Period 3
- MyDay, TruEye, Clariti 1day: Stenfilcon A contact lenses in Period 1, followed by narafilcon A contact lenses in Period 2 and somofilcon A contact lenses in Period 3
- MyDay, Clariti 1day, TruEye: Stenfilcon A contact lenses in Period 1, followed by somofilcon A contact lenses in Period 2 and narafilcon A contact lenses in Period 3
- Clariti 1day, TruEye, MyDay: Somofilcon A contact lenses in Period 1, followed by narafilcon A contact lenses in Period 2 and stenfilcon A contact lenses in Period 3
- Clariti 1day, MyDay, TruEye: Somofilcon A contact lenses in Period 1, followed by stenfilcon A contact lenses in Period 2 and narafilcon A contact lenses in Period 3
Period: First Wear Period (1 Day)
Arm/Group | TruEye, MyDay, Clariti 1day | TruEye, Clariti 1day, MyDay | MyDay, TruEye, Clariti 1day | MyDay, Clariti 1day, TruEye | Clariti 1day, TruEye, MyDay | Clariti 1day, MyDay, TruEye
Started | 4 | 4 | 4 | 4 | 4 | 4
Randomized and Treated | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Wear Period (1 Day)
Arm/Group | TruEye, MyDay, Clariti 1day | TruEye, Clariti 1day, MyDay | MyDay, TruEye, Clariti 1day | MyDay, Clariti 1day, TruEye | Clariti 1day, TruEye, MyDay | Clariti 1day, MyDay, TruEye
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Wear Period (1 Day)
Arm/Group | TruEye, MyDay, Clariti 1day | TruEye, Clariti 1day, MyDay | MyDay, TruEye, Clariti 1day | MyDay, Clariti 1day, TruEye | Clariti 1day, TruEye, MyDay | Clariti 1day, MyDay, TruEye
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat, defined as the set of all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | TruEye, MyDay, Clariti 1day | TruEye, Clariti 1day, MyDay | MyDay, TruEye, Clariti 1day | MyDay, Clariti 1day, TruEye | Clariti 1day, TruEye, MyDay | Clariti 1day, MyDay, TruEye | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (9.6) | 27.5 (4.0) | 33.0 (7.3) | 35.3 (4.6) | 26.3 (6.2) | 24.3 (2.4) | 30.0 (6.9)
Age, Customized [Number; unit: participants]
  18-64 years | 4 | 4 | 4 | 4 | 4 | 4 | 24
  ≥65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 2 | 4 | 2 | 15
  Male | 2 | 2 | 1 | 2 | 0 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Average Coefficient of Friction of Worn Lenses at 16 Hours
Description: Worn contact lenses were removed from the participant's eye and the coefficient of friction was measured by the inclined plane method. A lower coefficient of friction may indicate higher contact lens lubricity. The ex-vivo lubricity was carried out on one lens (one eye) only.
Time Frame: Day 1, Hour 16, each product
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- TruEye: Narafilcon A contact lenses worn for 16 hours in Period 1, Period 2, or Period 3
- MyDay: Stenfilcon A contact lenses worn for 16 hours in Period 1, Period 2, or Period 3
- Clariti 1day: Somofilcon A contact lenses worn for 16 hours in Period 1, Period 2, or Period 3
Arm/Group | TruEye | MyDay | Clariti 1day
Number analyzed (Participants) | 18 | 18 | 18
unitless | 0.0602 (0.00474) | 0.0576 (0.00338) | 0.0578 (0.00439)

2. Secondary Outcome: Average Coefficient of Friction of Unworn Lenses
Description: Unworn contact lenses were removed from the commercial packaging and the coefficient of friction of the unworn lenses was measured by the inclined plane method. A lower coefficient of friction may indicate higher contact lens lubricity.
Time Frame: Day 1 (each product)
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: unitless
Units Other Than Participants: contact lenses
Groups:
- TruEye: Narafilcon A contact lenses
- MyDay: Stenfilcon A contact lenses
- Clariti 1day: Somofilcon A contact lenses
Arm/Group | TruEye | MyDay | Clariti 1day
Number analyzed (Participants) | 18 | 18 | 18
Number analyzed (contact lenses) | 18 | 18 | 18
unitless | 0.0571 (0.00324) | 0.0571 (0.00260) | 0.0552 (0.00305)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study from the signing of informed consent (up to 17 days). This analysis population includes all participants exposed to investigational product.
Description: AEs were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs, whether or not related to the medical device, obtained through solicited and spontaneous comments from all exposed participants and reported based on the treatment received. Ocular AEs are presented for both eyes combined.
Groups:
- TruEye: Narafilcon A contact lenses worn bilaterally for 1 day (16 hours) in Period 1, Period 2, or Period 3
- MyDay: Stenfilcon A contact lenses worn bilaterally for 1 day (16 hours) in Period 1, Period 2, or Period 3
- Clariti 1day: Somofilcon A contact lenses worn bilaterally for 1 day (16 hours) in Period 1, Period 2, or Period 3
Arm/Group | TruEye | MyDay | Clariti 1day
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.